CLINICAL TRIAL: NCT03013803
Title: Acceptability Study on Nutricomp® Drink Plus Fibre in Adults
Acronym: Fuchsia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: B. Braun Melsungen AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HC-G-H-1610
Record Dates: First submitted 2016-12-19; First posted 2017-01-09 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-01

CONDITIONS: Adult Patients in Need of High-energy Oral Nutritional Supplementation
MeSH Terms: interventions — Dietary Fiber

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nutricomp Drink Plus Fibre (Experimental): Nutricomp® Drink Plus Fibre (flavours vanilla, coffee, peach-apricot and chocolate)
  Interventions: Dietary Supplement: Nutricomp Drink Plus Fibre

INTERVENTIONS:
Dietary Supplement: Nutricomp Drink Plus Fibre

SUMMARY:
Required for Advisory Committee for Borderline Substances (ACBS) approval. Aim of this study is to access the palatability, compliance and GI-tolerance of Nutricomp® Drink Plus Fibre to show that it is acceptable for patients in the United Kingdom.

ELIGIBILITY:
Inclusion criteria:

* Male and female participants ≥ 18 years of age
* Assessed to have malnutrition or be at risk of malnutrition by a Dietician within the investigator team. Assessment to include, but not limited to weight loss history, current BMI/MUST score, anamnesis, dietary intake history and predicted future oral intake.
* Anticipated period of nutritional support ≥ 12 days
* Patient has the capacity and is willing to provide informed consent.

Exclusion criteria:

* Participants with mental in capabilities who are unable to give informed consent
* Hypersensitivity to any of the active substances or excipients within the IP
* Severely impaired gastrointestinal function or complete failure
* More than 50% of nutrition from Parenteral Nutrition
* Simultaneous participation in another interventional study
* Participants who are unwilling or mentally and/or physically unable to adhere to study procedures
* Participants with dysphagia requiring thickened fluids
* Participants with significant renal impairment (CKD)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-12; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Occurrence of gastrointestinal tolerance parameters | Day 1 - day 13

SECONDARY OUTCOMES:
Occurrence of (further) adverse events during the treatment period (yes/no, if yes timing/duration/assumed cause/seriousness/severity) | Day 1 - day 13
Palatability evaluation performed under controlled condition using a questionnaire with a 5 point hedonic scale rang | Day 1 - day 13

CONTACTS AND LOCATIONS:
Locations (1):
- AC Health & Nutrition Ltd, Leigh-on-Sea, United Kingdom